CLINICAL TRIAL: NCT06913673
Title: Postoperative Pain and Incidence of Extrusion Following the Use of Two Intra-canal Medications in Retreatment of Single Rooted Teeth
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Ali, lecturer in endodontics, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1026/114
Record Dates: First submitted 2025-03-20; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Metapex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Metapex (Experimental): Non- surgical root canal retreatment with application of Metapex in to root canal after complete removal of the old obturation material.
  Interventions: Other: Metapex
- Group A:Bio-c Temp (Experimental): Non- surgical root canal retreatment with application of Bio-c Temp paste in to root canal after complete removal of the old obturation material.
  Interventions: Other: Bio-c Temp

INTERVENTIONS:
Other: Bio-c Temp — Intra-canal medication
  Arms: Group A:Bio-c Temp
Other: Metapex — Intra-canal medication
  Arms: Group A: Metapex

SUMMARY:
This study aims to compare the postoperative pain and incidence of extrusion of two intracanal medications in the retreatment of single-rooted teeth.

The main question it aims to answer is:

Does the injection of intra-canal medication into the shaped root canal after complete removal of the old obturating material lead to post-operative pain and paste extrusion to periapical tissues or not?

ELIGIBILITY:
Inclusion Criteria:

* Patients with failed endodontic treatment in single root teeth
* Systemic free

Exclusion Criteria:

* Muktirooted teeth

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of the post retreatment pain. | One week after re-treatment procdure
  Pain scores will be recorded on visual analog scale (VAS) using a 0 to 10 pain score basis with 0 being no pain and 10 being the worst pain the patient had ever experienced. (Record will be every 24h for 7 days)
Radiographic assessment of the extrusion of the paste into periapical tissues using Digital radiograph | Immediate after retreatment
  Extrusion of the paste into periapical incidence of extrusion: Conventional digital radiograph will be taken after using intracanal medication pastes.